CLINICAL TRIAL: NCT04824846
Title: An Interventional Study on Low Back Pain and Quality of Life Among the Ambulance Drivers in Malaysia's Hospitals
Brief Title: Low Back Pain and Quality of Life Among the Ambulance Drivers in Malaysia's Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ab Hamid Bin Abas, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-UD0020/18(R)
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain; Quality of Life
Keywords: LBP; QOL
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulance drivers with received Integrated back pain module (IBPM) (Experimental): Behavioral: Integrated back pain module (IBPM)
  Interventions: Behavioral: Integrated back pain module (IBPM)
- Ambulance drivers with received Health Educational Pamphlet. (Other): Other: Health Educational Pamphlet.
  Interventions: Other: Health Educational Pamphlet.

INTERVENTIONS:
Behavioral: Integrated back pain module (IBPM) — All Ambulance drivers will be screening with the Proforma to determine their low back pain symptoms. Those workers who are diagnosed with mechanical back pain during the 12 months fulfill a self-report quality of life questionnaire (SF-36). Then Integrated back pain module (IBPM) will be delivered to them after the introduction course conducted for 1 day and then the intervention will last for 6 months. Research staff will explain how to operate and use the module. Subjects must comply with all the care and prevention guidelines of the research module so that it achieves the expected results. They also need to complete the checklist provided in the Edmodo software via their respective smartphones.
  Arms: Ambulance drivers with received Integrated back pain module (IBPM)
Other: Health Educational Pamphlet. — In Health Educational Pamphlet (HEP) sessions, Participants will be taught the importance of movement and activity, pain management techniques, and methods for developing spinal posture awareness during activities of daily living (e.g., lifting, pushing, pulling, sitting, getting out of bed, and using a backpack).
  Arms: Ambulance drivers with received Health Educational Pamphlet.

SUMMARY:
The study is a community interventional study by using an integrated back pain module (IBPM). The purpose of this study is to find out if the module training has any benefit on Low Back pain among ambulance drivers. The effectiveness of the module is determined by baseline quality of life results compared with after the intervention program completed.

DETAILED DESCRIPTION:
An integrated back pain module (IBPM) will be implemented for ambulance drivers (Respondent) in peninsular Malaysia. Pre-intervention assessment and post-intervention assessment will be conducted in 18 government hospitals involved. There is nine Hospital in Perak that has been selected as an intervention group and nine Hospital in Kelantan will be the Control group. Two different regions are selected; the North region will be the intervention group (Perak) while East Coast will be the control group (Kelantan). The clinical benefits of the IBPM module low back pain and quality of life will be reported at the beginning and the end of the intervention and after a period of 6 months follow up.

The protocol for the intervention group (Perak) included five components of the education module (IBPM) such as the structure and function of the spine, causes of LBP, how to avoid low back pain at the workplace, Exercise methods, and psychology management. The overall objectives are to help ambulance driver manage their LBP and prevent future LBP recurrences. The first step of the protocol is subjects are required to attend an introductory course for one day and then the intervention will last for 6 months. Research staff will explain how to operate and use the module. Subjects must comply with all the care and prevention guidelines of the research module so that it achieves the expected results. They also need to complete the checklist provided in the Edmodo software via their respective smartphones. Tokens in the form of top-ups will be entered automatically after the checklist is received by researchers.

The exercise will be performed by participants 5 times per week for a total of 24 weeks. Each individual session will take around 5 minutes to perform exercises independently and sending their report through Edmodo. Light soft tissue exercises techniques such as active muscle stretching, and strengthening exercises will be used as needed to facilitate the educational module therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old.
* Working experience ≥ 1 year

Exclusion Criteria:

* Patients with Uncontrolled Chronic Illness such as Hypertension, Diabetes Mellitus, Osteoarthritis and Gout.
* Injury or surgery of the spine

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Ambulance Drivers in Malaysia's Hospitals
Enrollment: 198 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Quality of life in patients with Low back Pain before and after Integrated back pain module delivered. | Change from baseline, 6 weeks, 12 weeks, and 24 weeks
  Quality of life was assessed by Short-Form 36 Health Survey (SF-36) High scores indicate good quality of life and low scores represent poor quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Nazri B Shafei, Study Chair — University Science Malaysia
Locations (1):
- Ministry of Health Hospital, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No